CLINICAL TRIAL: NCT00111618
Title: An Open Label, Randomized, Phase II Study of AS1404 in Combination With Docetaxel in Patients With Hormone Refractory Metastatic Prostate Cancer
Brief Title: Study of AS1404 With Docetaxel in Patients With Hormone Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1404-203; NCT00119275 (obsolete NCT alias)
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Prostate Cancer
Keywords: vascular disrupting agent; safety; tolerability; efficacy; hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — vadimezan

INTERVENTIONS:
Drug: AS1404 (DMXAA)

SUMMARY:
The purpose of this trial is to confirm a safe dose of AS1404, to be given with docetaxel, and to see whether adding AS1404 and docetaxel together improves the outcome of the treatment, when compared to docetaxel alone.

DETAILED DESCRIPTION:
The overall aim of this study is to determine the safety, tolerability and efficacy of AS1404 in combination with docetaxel in patients with hormone refractory metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to, or greater than 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy greater than or equal to 3 months
* Histopathologically confirmed adenocarcinoma of the prostate
* Metastatic progressive androgen-independent prostate cancer with no previous chemotherapy treatment
* At least 4 weeks off of flutamide and 6 weeks off of bicalutamide and nilutamide
* Patients who have not undergone surgical castration must continue treatment with an luteinizing hormone-releasing hormone (LHRH) agonist. In those patients where, for some reason, the LHRH agonist has been discontinued prior to entry on the study, it should be reinstituted and disease progression must be documented.
* Hematological and biochemical indices at screening within the following ranges:

  * An absolute neutrophil count of greater than or equal to 1.5 x 10^9/L;
  * A platelet count of greater than or equal to 100 x 10^9/L;
  * A hemoglobin level of greater than or equal to 10 g/dL.
* Adequate hepatic and renal function, as defined by:

  * Serum bilirubin less than or equal to upper limit of normal (ULN);
  * SGOT and/or SGPT less than or equal to 1.5 x ULN concomitant with alkaline phosphatase less than or equal to 2.5 x ULN;
  * Serum creatinine less than or equal to 120 micromol/L or creatinine clearance greater than or equal to 60 mL/min.
* Be willing and able to provide written informed consent and, in the opinion of the Investigator, be able to comply with the study assessments and follow-up
* Serum testosterone no greater than 50 ng/mL (chemically castrated patients only)

Exclusion Criteria:

* Decreasing PSA levels after antiandrogen withdrawal
* Previous chemotherapy treatment for prostate cancer
* Patients who have received blood transfusions or growth factors to aid hematological recovery within two weeks of scheduled baseline visit
* Concurrent severe and/or uncontrolled co-morbid medical condition within 2 weeks of screening
* Previous exposure to AS1404 or other vascular targeting agents
* Clinically significant cardiac arrhythmias and known QTc prolongation (interval >450 msec)
* Evidence of severe or uncontrolled systemic disease that, in the opinion of the Investigator, might interfere with the patient's participation in the study
* A history of alcoholism; drug addiction; or any psychiatric condition, which, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures
* A history of hypersensitivity to taxanes or other drugs formulated with polysorbate 80
* Treatment with the following medications within two weeks of AS1404 administration or the expected need for such treatments during the study period:

  * Medications known to modulate serotonin;
  * Medications known to affect the QT interval;
  * Current treatment with, or the expected need during the treatment period for ketoconazole, erythromycin, troleandomycin, and/or cyclosporine. The use of other agents known to induce, inhibit, or that are metabolized by cytochrome P450-3A4 should be undertaken with caution.
* Concurrent or previous malignancy of a different tumor type within five years of starting the study, except for adequately treated non-melanoma skin cancer
* Clinical or radiological evidence of central nervous system (CNS) metastases
* Symptomatic peripheral neuropathy greater than or equal to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade II
* Evidence of any other significant clinical disorder or laboratory finding that, in the opinion of the Investigator, compromises the patient safety during study participation
* Participation in any prostate cancer investigational drug study in which the study drug has not subsequently obtained a product license
* Any other concurrent treatment for prostate cancer (with the exception of palliative radiotherapy) other than that specified in the protocol, including the use of herbal remedies, (e.g. saw palmetto)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Laboratory safety
Adverse event monitoring
Electrocardiogram (EKG)
Ophthalmic assessments
Tumor assessment
Time to progression and survival time
Prostate-specific antigen (PSA)
Pharmacokinetic sampling

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (27):
- United States (27):
  - Central Hematology Oncology Medical Group Inc, Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence Saint Joseph's Medical Center (PSJMC), Burbank, California
  - Pacific Oncology & Hematology Associates, Encinitas, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Clinical Research Unit, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, The Thomas and Dorothy Leavey Cancer Center, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Cancer Care Associates Medical Group, Inc, Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Stanford University Medical Center-Cancer Center, Stanford, California
  - University of Miami School of Medicine, Miami, Florida
  - Peachtree Hematology and Oncology, Atlanta, Georgia
  - Oncology Hematology Associates of Central Illinois,PC, Peoria, Illinois
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Staten Island Urological Research, Staten Island, New York
  - Biomedical Research Alliance of New York (BRANY), The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Virginia Health System, Charlottesville, Virginia
  - Marshfield Clinic Foundation, Marshfield, Wisconsin

REFERENCES:
- [Background] Jameson MB, Thompson PI, Baguley BC, Evans BD, Harvey VJ, Porter DJ, McCrystal MR, Small M, Bellenger K, Gumbrell L, Halbert GW, Kestell P; Phase I/II Trials Committee of Cancer Research UK. Clinical aspects of a phase I trial of 5,6-dimethylxanthenone-4-acetic acid (DMXAA), a novel antivascular agent. Br J Cancer. 2003 Jun 16;88(12):1844-50. doi: 10.1038/sj.bjc.6600992. PMID 12799625
- [Derived] Seshadri M, Spernyak JA, Maiery PG, Cheney RT, Mazurchuk R, Bellnier DA. Visualizing the acute effects of vascular-targeted therapy in vivo using intravital microscopy and magnetic resonance imaging: correlation with endothelial apoptosis, cytokine induction, and treatment outcome. Neoplasia. 2007 Feb;9(2):128-35. doi: 10.1593/neo.06748. PMID 17356709
- See also: Click here for additional information on Antisoma, the company sponsoring this study. — http://www.antisoma.com